CLINICAL TRIAL: NCT03466905
Title: Does Assessment of Ambulance Medical Service Leads to Reduced Number of Transports to the Emergency Room?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dalarna County Council, Sweden (Other)
Collaborators: County Council of Halland, Sweden (Other Government)
Responsible Party: Principal Investigator, Anneli Strömsöe, Registered Nurse, PhD, Dalarna County Council, Sweden
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Dnr 2016/393
Record Dates: First submitted 2017-02-12; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Emergency Medical Service; Assessment; Registered Nurse

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Intervention (Active Comparator): Assessment of Ambulance Medical Service
  Interventions: Other: Ambulant assessment
- Control (No Intervention): Local treatment guidelines

INTERVENTIONS:
Other: Ambulant assessment
  Arms: Intervention

SUMMARY:
There is a need to reduce the number of ambulance transports to the Emergency Room to the patients who are not in need of urgent medical care. There are currently no studies and the aim of the study is to investigate if the ambulance transports to the Emergency Room can be reduced by a dialogue between a Registered Nurse in ambulance and a Medical Doctor in the Primary Care (called "Ambulant assessment"). In this connection there is also a need to follow up patients that not have been transported to the Emergency Room, secondary ambulance transport, relapse within 48 hours, type of examination and treatment and mortality.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years
* ambulance missions in the Community of Borlänge/Falun (case) and Community of Leksand (control)
* weekday and weekend, 08:00 to 22:00
* initially evaluated not to need urgent Medical care according RETTS

Exclusion Criteria:

* initially evaluated need urgent Medical care according RETTS
* the patient unable to give consent to the study
* patient with existing care plan
* ambulance mission without patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11-07 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of visits to the Emergency Room | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- County Council of Dalarna, Falun, Dalarna County, Sweden